CLINICAL TRIAL: NCT01876446
Title: A Phase II Study of Single Agent Topoisomerase-I Inhibitor Polymer Conjugate, Etirinotecan Pegol (NKTR-102), in Patients With Relapsed Small Cell Lung Cancer
Brief Title: Pegylated Irinotecan NKTR 102 in Treating Patients With Relapsed Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Nektar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 225612; NCI-2013-01142 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 225612 (Other: Roswell Park Cancer Institute); P30CA016056 (NIH)
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Recurrent Small Cell Lung Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — etirinotecan pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (pegylated irinotecan NKTR 102) (Experimental): Patients receive pegylated irinotecan NKTR 102 IV over 90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Pegylated Irinotecan; Other: Pharmacological Study

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Pegylated Irinotecan — Given IV
  Other Names: NKTR 102; PEG-Irinotecan
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase II trial studies how well pegylated irinotecan NKTR 102 works in treating patients with small cell lung cancer that has returned after a period of improvement. Pegylated irinotecan NKTR 102 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the 18-week progression free survival (PFS) rate of relapsed small cell lung cancer (SCLC) patients treated with NKTR-102 (pegylated irinotecan NKTR 102).

SECONDARY OBJECTIVES:

I. To evaluate the objective response rate. II. To evaluate the duration of response. III. To evaluate the overall survival. IV. To evaluate the toxicity of NKTR-102 in this patient population.

TERTIARY OBJECTIVES:

I. To explore the correlation between UDP glucuronosyltransferase 1 family, polypeptide A cluster (UGTIA1) polymorphisms and NKTR-102 toxicities.

OUTLINE:

Patients receive pegylated irinotecan NKTR 102 intravenously (IV) over 90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent granted prior to initiation of any study-specific screening procedures, given with the understanding that the patient has the right to withdraw from the study at any time, without prejudice
* Histologic or cytologic diagnosis of SCLC (Note: patients with mixed histology are not eligible)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Presence of measurable disease defined as >= 1 lesion whose longest diameter can be accurately measured as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT)
* Previously treated SCLC with only one prior treatment regimen (cyclophosphamide/doxorubicin/vincristine [CAV] alternating with etoposide/cisplatin [EP] is acceptable)
* Resolution of all acute toxic effects of prior chemotherapy, radiotherapy, hormonal therapy, or surgery to National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 grade =< 1, except for diarrhea (which must be grade 0 without supportive antidiarrheal medications) and alopecia (any grade)
* Platelet count >= 100 x 10^9/L
* Hemoglobin (Hgb) >= 9 gm/dL
* Absolute neutrophil count (ANC) >= 1500/uL
* Serum creatinine =< 1.5 mg/dL or creatinine clearance > 45 mL/min; use either measured or calculated with Cockcroft-Gault formula
* Serum total bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 x ULN or =< 5 x ULN if caused by liver metastasis
* Women of childbearing potential must have a negative pregnancy test performed within seven days prior to the start of study drug; male and female subjects of child-bearing potential must agree to use double-barrier contraceptive measures, or avoidance of intercourse during the study and for 6 months after last investigational drug dose received

Exclusion Criteria:

* Previous anti-cancer chemotherapy, immunotherapy or investigational agents < 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to the first day of study defined treatment; palliative radiation < 2 weeks, biological therapy within 2 weeks, hormonal therapy within 1 week prior to day 1 cycle 1
* Prior treatment with a topoisomerase-I inhibitor (e.g., topotecan, irinotecan)
* Prior malignancy except for non-melanoma skin cancer and carcinoma in situ, unless diagnosed and definitively treated more than 5 years prior to enrollment
* Substance abuse, medical, psychological or social conditions that may, in the opinion of the Investigator, interfere with the patient's participation in the study or evaluation of the study results
* Known human immunodeficiency virus (HIV) infection
* Pregnancy or breast-feeding
* Concurrent administration or received cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inducers or inhibitors within 2 weeks prior to the first day of study drug treatment
* Patients with chronic or acute gastrointestinal (GI) disorders resulting in diarrhea of any severity grade; patients who are using chronic anti-diarrheal supportive care (more than 3 days/week) to control diarrhea in the 28 days prior to study entry
* Major surgery < 4 weeks or minor surgery (e.g. talc pleurodesis, excisional biopsy, etc) < 2 weeks prior to the first day of study defined treatment
* Have central nervous system (CNS) metastases (unless the patient has completed successful local therapy for CNS metastases and has been off corticosteroids for at least 4 weeks before starting study therapy); brain imaging is required in symptomatic patients to rule out brain metastases, but is not required in asymptomatic patients
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Unwilling or unable to follow protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-08-29 (Actual); Primary Completion 2017-07-18 (Actual); Study Completion 2020-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hongbin Chen, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (3):
- United States (3):
  - Roswell Park Cancer Institute, Buffalo, New York
  - Rochester General Hospital, Rochester, New York
  - Linden Oaks Medical Campus, Rochester, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- A: Chemo Resistant: Group A: chemo resistant - those progressing on first-line therapy < 3 months after completion of treatment.
  Treatment (pegylated irinotecan NKTR 102) Patients receive pegylated irinotecan NKTR 102 IV over 90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity
  Laboratory Biomarker Analysis: Correlative studies Pegylated Irinotecan: Given IV Pharmacological Study: Correlative studies
- B: Chemo Sensitive: Group B: chemo sensitive - those progressing on first-line therapy ≥ 3 months after completion of treatment.
  Treatment (pegylated irinotecan NKTR 102) Patients receive pegylated irinotecan NKTR 102 IV over 90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity
  Laboratory Biomarker Analysis: Correlative studies
  Pegylated Irinotecan: Given IV
  Pharmacological Study: Correlative studies
Period: Overall Study
Arm/Group | A: Chemo Resistant | B: Chemo Sensitive
Started | 20 | 18
Completed | 18 | 12
Not Completed | 2 | 6
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Physician Decision | 1 | 3

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Groups:
- Total: Total of all reporting groups
Arm/Group | A: Chemo Resistant | B: Chemo Sensitive | Total
Number analyzed (Participants) | 20 | 18 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 11 | 25
  >=65 years | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (8.7) | 61.9 (7.9) | 61.2 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 10 | 9 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 17 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
ECOG performance status [Count of Participants; unit: Participants] — ECOG Performance Status: Developed by the Eastern Cooperative Oncology Group GRADE 0 -Fully active, able to carry on all pre-disease performance without restriction, GRADE 1 -Restricted in physically strenuous activity but ambulatory and able to carry out work of light or sedentary nature, GRADE 2 -Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours, GRADE 3 -Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours, GRADE 4 -Completely disabled, GRADE 5 -Dead
  Participants
    Grade 0 | 9 | 8 | 17
    Grade 1 | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: 18 Week Progression-free Survival Rate
Description: The distribution of time to disease progression will be estimated in each group using the method of Kaplan-Meier at 18 weeks.
Time Frame: Time from registration to the date of first documented disease progression or death, assessed at 18 weeks
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A: Chemo Resistant | B: Chemo Sensitive
Number analyzed (Participants) | 20 | 18
percentage of participants | 35 [16 to 55] | 72 [46 to 87]

2. Secondary Outcome: Objective Tumor Response Measured With Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
Description: Objective tumor response will be tabulated overall (and by dose level if appropriate). Responses will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease in the cohorts (overall and by tumor group).
Time Frame: Up to 30 days
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A: Chemo Resistant | B: Chemo Sensitive
Number analyzed (Participants) | 20 | 18
percentage of participants | 20 [6 to 44] | 39 [17 to 64]

3. Secondary Outcome: Mean Duration of Response
Description: The mean duration of response for those participants that responded to treatment by arm.
Time Frame: Time from registration to death due to any cause, assessed up to 3 years
Population: All participants that responded to treatment
Measure: Mean (Standard Deviation); unit: months
Arm/Group | A: Chemo Resistant | B: Chemo Sensitive
Number analyzed (Participants) | 4 | 7
months | 5.4 (3.8) | 7.0 (6.8)

4. Secondary Outcome: Best Response
Description: Count of participants by best response, defined as best objective status recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since treatment started), measured by RECIST 1.1
  Tumor response is defined as a complete response (CR) or partial response (PR) by RECIST 1.1 criteria, which will be evaluated by CT scan every other cycle. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT scan: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 30 days
Population: All treated and eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | A: Chemo Resistant | B: Chemo Sensitive
Number analyzed (Participants) | 20 | 18
Participants
  CR Complete Response/Remission | 0 | 1
  PR Partial Response/Remission | 4 | 6
  SD Stable Disease | 6 | 7
  PD Progressive Disease | 9 | 2
  NE Not Evaluable | 1 | 2

5. Secondary Outcome: Median Overall Survival
Description: The distribution of survival time was be estimated in each group using the method of Kaplan-Meier.
Time Frame: Time from registration to death due to any cause, assessed up to 3 years
Population: All treated and eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A: Chemo Resistant | B: Chemo Sensitive
Number analyzed (Participants) | 20 | 18
months | 7.4 [2.9 to 11.7] | 7.1 [4.8 to 14.7]

6. Secondary Outcome: Incidence of Adverse Events, Assessed Using NCI CTCAE v 4.0
Description: Count of participants by maximum graded according to NCI CTCAE v 4.0 of any adverse event by arm.
  Please refer to the adverse event reporting for more detail.
Time Frame: Up to 30 days
Population: All treated and eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | A: Chemo Resistant | B: Chemo Sensitive
Number analyzed (Participants) | 20 | 18
Participants
  Grade 1 | 7 | 1
  Grade 2 | 3 | 6
  Grade 3 | 9 | 9
  Grade 4 | 0 | 1
  Grade 5 | 0 | 1
  Grade 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: From time of Cycle 1 Day 1 until 30 days after receiving last dose of study drug, an average of 4 months (range 1 to 21 months).
Arm/Group | A: Chemo Resistant | B: Chemo Sensitive
All-Cause Mortality (participants affected / at risk) | 0/20 | 1/18
Serious Adverse Events (participants affected / at risk) | 4/20 | 4/18
Other Adverse Events (participants affected / at risk) | 19/20 | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Chemo Resistant (N=20) | B: Chemo Sensitive (N=18)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (4) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Chemo Resistant (N=20) | B: Chemo Sensitive (N=18)
Anaemia (Blood and lymphatic system disorders) | 5 (9) | 3 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1)
Photopsia (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (2) | 3 (10)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 4 (7)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (6)
Diarrhoea (Gastrointestinal disorders) | 10 (25) | 12 (33)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 1 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (13) | 10 (16)
Retching (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (10) | 5 (13)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 7 (13) | 7 (11)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 1 (1)
Oedema (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (2)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Candidiasis (Infections and infestations) | 0 (0) | 1 (2)
Pelvic abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase (Investigations) | 0 (0) | 2 (4)
Blood alkaline phosphatase (Investigations) | 0 (0) | 1 (2)
Blood creatinine (Investigations) | 1 (4) | 0 (0)
Haemoglobin (Investigations) | 1 (6) | 4 (6)
Lymphocyte count decreased (Investigations) | 4 (9) | 4 (9)
Neutrophil count decreased (Investigations) | 4 (15) | 2 (2)
Platelet count decreased (Investigations) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 7 (9) | 4 (5)
White blood cell count decreased (Investigations) | 6 (21) | 3 (6)
Decreased appetite (Metabolism and nutrition disorders) | 3 (4) | 7 (12)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (4) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (4) | 4 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Amputation stump pain (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 3 (6)
Dysgeusia (Nervous system disorders) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (2)
Hallucination (Psychiatric disorders) | 0 (0) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0)
Vasodilatation (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-27): https://cdn.clinicaltrials.gov/large-docs/46/NCT01876446/Prot_SAP_000.pdf